CLINICAL TRIAL: NCT06057727
Title: BE IMMUNE: Behavioral Economics to IMprove and Motivate Vaccination Using Nudges Through the EHR
Brief Title: Behavioral Economics to Improve Flu Vaccination Using EHR Nudges
Acronym: BE IMMUNE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Washington (Other)
Responsible Party: Principal Investigator, Shivan J Mehta, Associate Chief Innovation Officer, Associate Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 851838; R33AG068945 (NIH)
Record Dates: First submitted 2023-09-18; First posted 2023-09-28 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Behavior, Health; Flu; Flu Vaccination
Keywords: Flu Vaccine Uptake; EHR Nudge; Behavioral Economics; Health Disparities
MeSH Terms: conditions — Health Behavior; Influenza, Human

STUDY DESIGN:
Intervention Model Description: We will randomize primary care clinics 2:1 to the intervention arm or control arm using covariate-constrained randomization. Patients identified as at high-risk for non-completion of the flu vaccine will be additionally randomized 1:1 at the individual level to receive an additional intensification nudge compared with the multi-component nudge intervention alone.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Clinics randomized to the control arm will receive standard of care.
- Intervention Arm (Experimental): Clinics randomized to the intervention arm will receive the toolkit of clinician and patient facing nudges. Patient nudges will be pre-visit text message reminders (standard messaging content). Clinician nudges will be monthly peer comparison feedback and default pended orders.
  Interventions: Behavioral: Pre-visit patient text messaging; Behavioral: Default pended order; Behavioral: Monthly peer comparison feedback
- High Risk Intensification Arm (Experimental): Patients in the intervention clinics identified as high risk for noncompletion of the flu vaccine will be randomized 1:1 to receive the high risk intensification arm or remain in the standard intervention arm. Patients in the high risk intensification arm will receive an additional bidirectional texting component.
  Interventions: Behavioral: Pre-visit patient text messaging; Behavioral: Default pended order; Behavioral: Monthly peer comparison feedback; Behavioral: High risk bidirectional pre-visit text messaging

INTERVENTIONS:
Behavioral: Pre-visit patient text messaging — Patients will be sent text message reminders 3 days and 24 hours prior to their scheduled primary care visit. The messages will inform the patient that a flu shot has been reserved for them at their upcoming appointment and encouraging the patient to ask their provider about receiving the vaccine.
  Arms: High Risk Intensification Arm; Intervention Arm
Behavioral: Default pended order — A default pended order for the flu vaccine will be pended to the patient's upcoming primary care encounter and will be visible to the provider during the visit encounter. Clinical staff will have the option of signing the order or dismissing it if they deem it inappropriate for a given patient.
  Arms: High Risk Intensification Arm; Intervention Arm
Behavioral: Monthly peer comparison feedback — Each month, clinicians will be sent an email containing what percent of their eligible patients received the flu vaccine and how that compares to other peer clinicians in the intervention.
  Arms: High Risk Intensification Arm; Intervention Arm
Behavioral: High risk bidirectional pre-visit text messaging — High risk patients randomized to receive the high risk intensification nudge will receive a bidirectional text messaging component prior to their visit. This intervention will query the patient about common questions or concerns about receiving the flu vaccine. If the patient responds, it will provide additional educational materials based on the patient's specific concern(s).
  Arms: High Risk Intensification Arm

SUMMARY:
This study will be a multisite, cluster randomized, pragmatic trial to evaluate the effectiveness of personalized nudges to clinicians and patients, relative to a control, to increase flu vaccination rates among older adults in accordance with CDC guidelines. This will include clinician and patient level nudge interventions, with an additional, intensified nudge intervention for patients identified as high risk for not receiving a flu vaccine. Among the intervention clinics, patients will receive pre-visit text message reminders about the flu vaccine, and clinicians will receive a default pended order in the visit encounter in the EHR, along with monthly peer comparison feedback about their flu vaccine completion rate. Patients identified as high risk for noncompletion will be individually randomized to receive an additional bidirectional text message nudge or the standard text messaging.

DETAILED DESCRIPTION:
Many older adults are at risk of illness, hospitalization, and death from vaccine-preventable diseases. More than half of older adults in the United States are not vaccinated for flu which has remained relatively constant over the past decade, and there are racial, ethnic, and socioeconomic disparities in care. In this study, we will evaluate personalized nudges to clinicians and patients to help increase flu vaccination rates during primary care visits among older adults, with a particular focus on population subgroups at high risk for vaccine noncompletion. In a partnership between Penn Medicine and University of Washington (UW) Medicine, this will be a 6-month, multisite, cluster randomized, pragmatic trial with an additional intensification arm for high-risk patients.

ELIGIBILITY:
Patient Inclusion Criteria:

All patients must meet the following criteria to be eligible:

1. Age >50 years
2. A scheduled new or return (non-urgent/sick) primary care appointment at one of the study practices at the Penn Medicine, UW Medicine, or Lancaster General Hospital
3. Have not received their annual flu vaccine during the active intervention period (September- February)
4. Eligible to receive the flu vaccine

For the high risk intensification nudge, at least one of the following criteria must be met to be considered high risk and randomized to receive the intensification nudge:

1. Age ≥ 70 years
2. Living in a lower income community (lowest quartile, zip-code based)
3. Did not receive a flu vaccine in the previous calendar year
4. Self-identifies as Non-Hispanic Black

Patient Exclusion Criteria:

1. Have a documented allergy to flu vaccine
2. Have a flu vaccine exclusion modifier in Health Maintenance
3. Have opted out of research according to individual site guidelines and policies
4. Have no phone number (home or mobile) listed in their chart

Clinician Inclusion Criteria:

Clinicians must meet the following criteria to be eligible to receive peer comparison feedback:

1. Practicing physician (MD, DO) or advanced practice provider (NP, PA) with the exception of residents and fellows
2. Have a minimum patient panel of at least 50 patients, and
3. Practicing at a clinical site randomized to receive the clinic-level nudge interventions.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80039 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD,MBA,MSHP, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
We will share our analytical code(s).
Supporting Information: Study Protocol, Analytic Code
Time Frame: Within one year of trial completion
Access Criteria: All inquiries related to the code should be directed to the PI.

REFERENCES:
- [Derived] Mehta SJ, Waddell KJ, Linn KA, Brophy C, Liang J, Park SH, Reitz C, Williams K, Couzens C, Staloff J, White AA, Rhodes C, Liao JM, Navathe AS. Nudges to Clinicians and Patients for Influenza Vaccines During Visits: The BE IMMUNE Randomized Clinical Trial. JAMA Intern Med. 2026 Jan 5:e257133. doi: 10.1001/jamainternmed.2025.7133. Online ahead of print. PMID 41490010
- [Derived] Waddell K, Mehta SJ, Navathe A, Linn K, Park SH, White A, Staloff J, Rhodes C, Couzens C, Goel K, McDonald C, Reitz C, Williams K, Liao JM. Behavioural economics to improve and motivate vaccination in primary care using nudges through the electronic health record: rationale and design of the BE IMMUNE randomised clinical trial. BMJ Open. 2024 Nov 18;14(11):e086698. doi: 10.1136/bmjopen-2024-086698. PMID 39557547

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Waiver of informed consent obtained. Patients were identified via Epic Clarity Query 4 days prior to their eligible primary care visit between September 25, 2023 - February 20, 2024. Patients were only counted once within the study window at their first primary care visit. Total protocol enrollment: 80,039 patients.
Pre-assignment Details: Clinics were randomized 2:1 to intervention and control. Patients seen at an intervention clinic and identified as high risk were further randomized 1:1 to standard messaging or an intensification nudge. The high risk individual randomization is nested within the intervention arm resulting in an overlap of patients where high risk individuals (41,909 of the 52,526) contribute both to estimation of the overall intervention effect and comparison of text messaging intensity among high risk patients
Units Other Than Participants: Clinics
Groups:
- Control: Patients in clinics randomized to the control arm will receive standard of care.
- Intervention: Patients in clinics randomized to the intervention arm will receive the toolkit of clinician and patient facing nudges. Patient nudges will be pre-visit text message reminders (standard messaging content). Clinician nudges will be monthly peer comparison feedback and default pended orders.
- High Risk - Standard Messaging: Patients in the intervention clinics identified as high risk for noncompletion of the flu vaccine were randomized 1:1 to receive the high risk intensification messaging or remain in the standard messaging arm. Patients in the high risk standard messaging arm received the same standard messaging as average risk patients.
- High Risk - Intensification Messaging: Patients in the intervention clinics identified as high risk for noncompletion of the flu vaccine were randomized 1:1 to receive the high risk intensification messaging or remain in the standard messaging arm. Patients in the high risk intensification group received an additional bidirectional texting component in addition to the standard messaging.
- High Risk - Not Individually Randomized: Patients in the intervention clinics identified as high risk for noncompletion of the flu vaccine who were not individually randomized as a result of an automation issue. These patients still received the clinician nudges (default pended orders and peer comparison feedback) but did not receive any standard or intensification messaging.
Period: Clinic Level Randomization
Arm/Group | Control | Intervention | High Risk - Standard Messaging | High Risk - Intensification Messaging | High Risk - Not Individually Randomized
Started | 27513; 16 Clinics | 52526; 32 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Completed | 27513; 16 Clinics | 52526; 31 Clinics (1 primary care clinic resulted in no patients due to a change in the department ID code that was not reflected in the enrollment query) | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Not Completed | 0; 0 Clinics | 0; 1 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Individual Level Randomization
Arm/Group | Control | Intervention | High Risk - Standard Messaging | High Risk - Intensification Messaging | High Risk - Not Individually Randomized
Started | 0; 0 Clinics | 0; 0 Clinics | 20440; 0 Clinics (A subset of the 52,526 patients seen at intervention clinics who are identified as high risk and then individually randomized to receive standard messaging.) | 20412; 0 Clinics (A subset of the 52,526 patients seen at intervention clinics who are identified as high risk and then individually randomized to receive intensification messaging.) | 1057; 0 Clinics (A subset of the 52,526 patients seen at intervention clinics who are identified as high risk but were not individually randomized. Received no messaging.)
Completed | 0; 0 Clinics | 0; 0 Clinics | 20440; 0 Clinics | 20412; 0 Clinics | 1057; 0 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for the Main Study Period only - Clinic Level Randomization (Control and Intervention). Patients in the High Risk arms are accounted for in the Intervention arm as a whole, but were additionally randomized at the Individual Level, as noted in the Participant Flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 27513 | 52526 | 80039
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (10.0) | 66.1 (10.3) | 65.8 (10.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 12128 | 22747 | 34875
  Female | 15162 | 29640 | 44802
  Unknown | 223 | 139 | 362
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 138 | 266 | 404
  Asian | 2167 | 3412 | 5579
  Native Hawaiian or Other Pacific Islander | 135 | 144 | 279
  Black or African American | 6767 | 11928 | 18695
  White | 16534 | 33638 | 50172
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1772 | 3138 | 4910
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino/ Unknown | 26161 | 50733 | 76894
  Ethnicity: Hispanic or Latino | 1352 | 1793 | 3145
Lowest Quartile Income by Zip Code [Count of Participants; unit: Participants]
  Above Lowest Income Quartile by Zip Code | 19406 | 37064 | 56470
  Lowest Income Quartile by Zip Code | 8107 | 15462 | 23569

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Receive the Flu Vaccine at the Visit
Description: The primary outcome is flu vaccination completion during the first eligible primary care visit.
Time Frame: 4 days from enrollment, at the eligible visit
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention | High Risk - Standard Messaging | High Risk - Intensification Messaging | High Risk - Not Individually Randomized
Number analyzed (Participants) | 27513 | 52526 | 20440 | 20412 | 1057
Participants | 7305 | 16663 | 6142 | 6142 | 312

2. Secondary Outcome: Proportion of Patients Who Receive the Flu Vaccine Within 3 Months After the Visit
Description: The secondary outcome is flu vaccination completion within 3 months after the first eligible primary care visit.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention | High Risk - Standard Messaging | High Risk - Intensification Messaging | High Risk - Not Individually Randomized
Number analyzed (Participants) | 27513 | 52526 | 20440 | 20412 | 1057
Participants | 9371 | 19892 | 7329 | 7371 | 385

ADVERSE EVENTS:
Time Frame: Each patient was monitored for adverse events for 3 months. Adverse events were collected mid-way through the trial at 3 months for all participants enrolled through the end of December 2023 and again at the end of the trial follow up period, 3 months after enrollment ended (May 2024), for all enrolled participants.
Description: Per our DSMB-approved DSMP, severe adverse events will not include death as no reasonable evidence exists to suggest death would result from outreach or communication to encourage standard clinical care for flu vaccination. Therefore, All-Cause Mortality was not assessed. Adverse events are assessed for the Main Study Period arms only - Control (except Messaging, see footnote) and Intervention - as the patients in the High Risk arms are already accounted for in the Intervention arm total.
Groups:
- Intervention: Patients in clinics randomized to the intervention arm will receive the toolkit of clinician and patient facing nudges. Patient nudges will be pre-visit text message reminders (standard messaging content). Clinician nudges will be monthly peer comparison feedback and default pended orders. Includes all intervention arm patients, including high risk.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/27513 | 1/52526
Other Adverse Events (participants affected / at risk) | 5/27513 | 817/52526
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=27513) | Intervention (N=52526)
Flu Vaccine Reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Reaction requiring emergency department or hospital care.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Control (N=27513) | Intervention (N=52526)
Messaging Opt-out (Social circumstances) | 0/0 (0) | 795 (795) — Patient frustration with messaging or outreach. Messaging opt-out was not assessed for control patients as they did not receive any messaging.
Duplicate Vaccination (Surgical and medical procedures) | 5 (5) | 22 (22) — Duplicate flu vaccination within the recommended interval.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-10-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT06057727/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT06057727/SAP_001.pdf